CLINICAL TRIAL: NCT04915014
Title: Prospective Multicentric Randomized Trial Comparing the Efficacy and Safety of Sleeve Gastrectomy With Transit Bipartition (SG+TB) Versus Roux-en-Y Gastric Bypass (RYGB)
Brief Title: Sleeve Gastrectomy With Transit Bipartition(SG+TB) Versus Roux-en-Y Gastric Bypass (RYGB) for Type 3 Obesity
Acronym: BIPASS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020_10; 2020-A02656-33 (Other: ID-RCB number,ANSM); PHRC-19-031 (Other: DGOS number, PHRC-N)
Record Dates: First submitted 2021-05-19; First posted 2021-06-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Severe Obesity
Keywords: Severe obesity; Type 2 diabetes; Metabolic syndrome; Surgery; Malnutrition
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2; Metabolic Syndrome; Malnutrition | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic sleeve gastrectomy with transit bipartition (SG +TB) (Experimental): One arm benefiting from a laparoscopic sleeve gastrectomy with transit bipartition (SG +TB)
  Interventions: Procedure: sleeve gastrectomy with transit bipartition (SG +TB)
- laparoscopic Roux-en-Y gastric bypass (RYGB) (Sham Comparator): One arm benefiting from a laparoscopic Roux-en-Y gastric bypass (RYGB)
  Interventions: Procedure: Roux-en-Y gastric bypass (RYGB)

INTERVENTIONS:
Procedure: sleeve gastrectomy with transit bipartition (SG +TB) — In case of a first intention procedure, a typical sleeve gastrectomy is performed, calibrated on a 36 French bougie, stapling starting 4 to 6 cm from the pylorus. Antecolic gastroileal anastomosis is performed 250 cm from the ileocecal transition, on the antrum using a linear stapler (45-mm gold cartridge) or hand-sewn (at least 3 cm wide on the stomach). Laterolateral enteroanastomosis is performed 120 cm from the ileocecal junction. Thus, alimentary limb is 130cm and common limb 120cm.
  Arms: laparoscopic sleeve gastrectomy with transit bipartition (SG +TB)
Procedure: Roux-en-Y gastric bypass (RYGB) — A small gastric pouch (30 cc) is performed. Antecolic gastroileal anastomosis is performed 200 cm from the Treitz junction, using a linear stapler (45-mm gold cartridge) or hand-sewn (at least 3 cm wide on the stomach). Laterolateral enteroanastomosis is performed 50 cm from the Treitz junction. Thus, alimentary limb is 150cm and biliary limb 50cm.
  Arms: laparoscopic Roux-en-Y gastric bypass (RYGB)

SUMMARY:
Obesity is a major public health problem worldwide. Bariatric surgery has proved to be the most effective treatment of morbid obesity in terms of weight reduction and remission of co-morbid conditions during long-term follow-up. Sleeve Gastrectomy (SG) has become the most performed intervention either worldwide or in France, where SG represents more than 60% of bariatric interventions and 114,817 patients operated between 2013 and 2016.

Maximum Excess weight loss (%EWL) after SG is obtained at one-year post surgery. Then it has been largely reported in the literature that patients could present mild, moderate or important (notably in the super obese patients) weight regain associated with comorbidity relapse motivating redo surgery. Like in revisional surgery, operating super-obese patient (BMI ≥50 kg/m2) is a challenge. It has been shown that achieving significant weight loss was more difficult in patients with a BMI ≥ 50 compared to lower BMIs.

DETAILED DESCRIPTION:
In these 2 populations of patients, more malabsorptive procedures like long limb One Anastomosis Gastric Bypass or Bilio-Pancreatic Diversion with Duodenal Switch could be more efficient but induce technical difficulties (high complication rate) and can be responsible for malnutrition (vitamin deficiencies, hypoalbuminemia…). That's why, in case of revisional surgery or for high BMI patients,laparoscopic Roux-en-Y gastric bypass (RYGBP) is still considered as the gold standard and is the most performed intervention. To obtain better weight loss safely,Santoro et al. promoted the sleeve gastrectomy with transit bipartition (SG+TB), a new intervention coupling a SG without interrupting pathway through the duodenum and preserving the pylorus and a long biliary limb RYGBP.

Hypothesis: Because there is no duodenal and jejunal exclusion, malnutrition is expected to be less frequent after SG+TB compared to BPD/DS. Its anastomosis on the antrum makes SG+TB easier to perform in super-obese patient than standard RYGB but more efficient in term of weight loss. Compared to BPD/DS or SADI which involves dissection of the duodenum and the confection of a duodenojejunostomy, SG+TB is also expected to be easier then safer.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has benefited from a pluridisciplinary evaluation, with a favorable opinion for SG+TB or RYGB as a first intention procedure with BMI ≥40 kg/m2 or BMI ≥ 35 kg/m2 associated with one co-morbidity which will be improved by surgery (according to HAS 2009 recommendation3) OR as a second intention procedure (revisional surgery) after failure of Sleeve gastrectomy (defined as insufficient weight loss at 18 months after surgery (EWL% <50), or as weight regain (+ 20%)).
* Patient who had benefited from an Upper GI Endoscopy with biopsies to look for Helicobacter Pylori (HP) and a HP eradication.
* Patient who understands and accepts the need for a long-term follow-up
* Patient who agrees to be included in the study and who signs the informed consent form
* Patient affiliated to a healthcare insurance plan

Exclusion Criteria:

* History of previous bariatric surgery, other than a Sleeve Gastrectomy
* Patient with current BMI > 60 kg/m2
* Presence of a severe and evolutive life threatening pathology, unrelated to obesity
* History of Chronic inflammatory bowel disease
* Type 1 Diabetes
* Pregnancy or desire to be pregnant during the study
* Nursing woman
* Presence of Pylori Helicobacter resistant to medical treatment
* Presence of a non-healed gastro-duodenal ulcer or diagnosed less than 2 months previously
* Severe esophagitis (grade C of Los Angeles classification)
* Hiatal hernia
* Patients with unstable psychiatric disorder, under supervision or guardianship
* Patient who does not understand French/ is unable to give consent
* Patient not affiliated to a French or European healthcare insurance
* Patient who has already been included in a trial which has a conflict of interests with the present study
* Patient incarcerated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The Excess Weight Loss percentage (EWL%) | at 2 years after surgery
  The Excess Weight Loss percentage (EWL%) calculated with the following formula: ((weight at 2 years visit - initial weight (kg)) / (initial weight - ideal weight)) X 100 Ideal weight defined as the weight corresponding to a BMI = 25 kg/m2. Initial weight defined as preoperative weight at V1. All weights are expressed in kg

SECONDARY OUTCOMES:
Change nutritional status assessment | from baseline (before surgery) to 24 months after surgery
  Nutritional profil : Hemoglobin (g/l), albumin (g/l), prealbumin (g/l)
Change in liver status assessment | from baseline (before surgery) to 24 months after surgery
  Liver parameters ( ALT AST GGT Alkaline phosphatases, Total bilirubin, prothrombin time, urea, creatininemia concentration)
Change in vitamins status assessment | from baseline (before surgery) to 24 months after surgery
  vitamins profil (vitamin A B1, B6 B9, B12, C , D and E concentration)
Change in mineral status assessment | from baseline (before surgery) to 24 months after surgery
  Mineral profil ( ferritin, potassium, calcium,iron, transferrin, magnesium, selenium, zinc phophore concentration)
24-hour steatorrhea quantified at 6 months | At 6 months
  24-hour steatorrhea is assessed to evaluate denutrition, expressed in g of lipid/24hr
Evolution of muscle mass assessed by bioelectrical impedance analysis | from baseline to 24 months after surgery
  muscle mass is assessed to evaluate denutrition.
Evolution of muscle mass assessed by grip strength test. | from baseline to 24 months after surgery
  muscle mass is assessed to evaluate denutrition.
Complications rate within 2 years according to Dindo-Clavien classification | within 2 years
  complications rate is assessed to evaluate safety of the procedure
Length of hospital stay defined as the number of days of hospitalization | up to 2 week
  length of hospital stay for the surgical procedure
Evolution from baseline to 24 months after surgery of HbA1c level, HDL, LDL and triglycerides | from baseline to 24 months after surgery
  Evolution from baseline to 24 months after surgery of HbA1c level (expressed in %), fasting glycemia (expressed in mmol/l or g/l), HDL (expressed in mmol/l or g/l), LDL (expressed in mmol/l or g/l) and triglycerides (expressed in mmol/l)
Evolution from baseline to 24 months of insulinoresistance defined by HOMA-IR calculated with fasting blood glucose and fasting insulinemia12 | from baseline to 24 months
  assessment of insulinoresistance
Change of the GIQLI score | from baseline to 24 months after surgery
  This questionnaire consists of 36 items exploring 5 dimensions or subscales: symptoms, physical condition, emotions, social integration and the effect of any medical treatment. For each item, 5 responses will be proposed to patients and for each answer, a score is assigned, ranging from 0 to 4 (highest score = 144). A high score defines a more favorable health state
Change of the SF36 scores | from baseline to 24 months after surgery
  This questionnaire taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.
Change in Sigstad questionnaire score (dumping syndrome). | from baseline to 24 months after surgery
  The Sigstad questionnaire allows the identification and diagnosis of postoperative hypoglycemia: a score > 7 suggests a dumping and a score <4 suggests another diagnosis.
  Complementary questions regarding timing of dumping (<30 min or >1h30) will be asked if Sigstad score >7.
Change of food choices and preferences assessed by the Leeds Food Preference Questionnaire (LFPQ) score. | from baseline to 24 months after surgery
  The Leeds Food Preference Questionnaire provides measures of different components of food preference and food reward. Participants are presented with an array of pictures of individual food items common in the diet. Foods in the array are chosen by the experimenter from a validated database to be either predominantly high (>50% energy) or low (<20% energy) in fat but similar in familiarity, protein content, sweet or non-sweet taste and palatability. Outcome measured are explicit Liking, explicit wanting, implicit wanting and food choice.
  Scores for explicit liking and explicit wanting range from 0-100 with a typical mean (±S.D.) of 60±18 Scores for Food Choice range from 0-48 and have a typical mean of 24±10 or for the appeal bias range from -48-48 with a typical mean of -5±15.
  Scores for Implicit Wanting typically range from -100-100 (due to RT there is no fixed min-max value) and have a typical mean of ±10±25 or for the appeal bias a typical mean of -10±30.
Change of physical activity assessed by the International Physical Activity Index (IPAQ) score. | from baseline to 24 months after surgery
  The International Physical Activity Questionnaire assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives to estimate total physical activity in MET-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Robert CAIAZZO, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (8):
- France (8):
  - Hop Claude Huriez Chu Lille, Lille
  - CHU de Lyon, Lyon
  - CHU de Nantes, Nantes
  - CHU Orléans, Orléans
  - AP-HP Hôpital Bichat, Paris
  - AP-HP Hôpital Georges Pompidou, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Nancy, Vandœuvre-lès-Nancy